CLINICAL TRIAL: NCT01101607
Title: Closed Reduction and Cast Immobilization of Distal Radius Fractures by Pediatric Emergency Medicine
Brief Title: Closed Reduction of Distal Forearm Fractures by Pediatric Emergency Medicine Physicians: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMotion Orthopaedic Research Center (Other)
Collaborators: University of Tennessee (Other); Le Bonheur Children's Hospital (Other); Campbell Clinic (Other)
Responsible Party: Dick Tarr, InMotion Orthopaedic Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MHIRB 2008-006
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Pediatric Distal Forearm Fractures
Keywords: Pediatrics; Distal Forearm fractures; Pediatric Emergency Medicine; Pediatric Orthopedics
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pediatric Emergency Physician (Active Comparator): Patients randomized to Pediatric Emergency Physician Group will have their fracture reduced by a Pediatric Emergency Physician
  Interventions: Procedure: Distal Forearm Fracture Reduction
- Orthopaedic physician (Active Comparator): Patients to be randomized to Orthopaedic physician Group will have their fracture reduced by an Orthopaedic Physician
  Interventions: Procedure: Distal Forearm Fracture Reduction

INTERVENTIONS:
Procedure: Distal Forearm Fracture Reduction — Fracture reduction

SUMMARY:
Distal forearm fractures are amongst the most frequently encountered orthopedic injuries in the pediatric emergency department (ED). Immediate closed manipulation and cast immobilization, is still the mainstay of management. The initial management of non-displaced or minimally displaced extremity fractures and relocation of uncomplicated joint dislocations is part of the usual practice of emergency medicine. Although focused training in fracture-dislocation reduction techniques is a part of the core curriculum of emergency medicine training programs, there is limited data discussing outcomes following restorative fracture care by pediatric emergency medicine (PEM)physicians.

The primary objective of this study is to compare length-of-stay and clinical outcomes after closed manipulation of uncomplicated, isolated, distal forearm fractures, by PEMs to those after manipulation by pediatric orthopedic surgeons. Our hypothesis is that there is no difference in emergency department length-of-stay when fracture reduction is performed by a PEM versus a post graduate year 3 or 4 orthopedic resident. Secondary outcomes that will be assessed include: loss of reduction needing re-manipulation at follow up, cast related complications, radiographic and functional healing at 6-8 weeks post injury.

DETAILED DESCRIPTION:
Pediatric forearm fractures are common injuries and a frequent cause for an emergency room admission. Ward et al have outlined the demands that emergency department coverage places on practicing orthopedic surgeons. Assuming no statistically significant differences in outcomes, there are potential advantages of having PEMs provide restorative fracture care at the initial visit. This practice would permit judicious orthopedic consultation at a time when several emergency department's are facing an "on call" specialist coverage crisis and there exists a nationwide shortage of fellowship trained pediatric orthopedic specialists, in addition to ACGME mandated duty hour restrictions for orthopedic residents.

Pershad et al conducted a retrospective study with historical controls, of 60 patients with distal radius fracture that were reduced by an orthopedic resident or PEM physician. In this review, there were no differences in rates of re-intervention to restore fracture alignment or ED length-of-stay between the two groups.Mean facility charges were lower in the group treated by PEMs.

It is our hypothesis that with goal directed training, PEM physicians can perform closed reduction of uncomplicated distal forearm fractures with outcomes that are similar to when fracture reduction is performed by senior orthopedic resident physicians.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will include patients who present to LeBonheur Emergency room with an angulated or displaced distal radius fracture that meet standard orthopaedic criteria for manipulation. Distal forearm will be defined anatomically as the distal third of the radius or ulna.

Exclusion Criteria:

The exclusion criteria will be patients with an open fracture, neurovascular compromise at presentation or who have undergone prior manipulation of their fracture. Prior manipulation of a fracture is defined when a patient has their fracture manipulated at an outlying facility prior to arriving to LeBonhuer emergency room.

-

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Adequate Alignment of the forearm fracture | 5-7 days post-injury
  The primary outcome in this study is the determination of whether there is adequate alignment of the fracture at 5-7 days post-injury. The proportion of patients with adequate alignments will be compared between the Pediatric Emergency Medicine and the Orthopaedic groups.

SECONDARY OUTCOMES:
Complications | 6-8 weeks post-injury
  Secondary outcomes to be assessed include incidence of failed apposition needing remanipulation at follow-up, cast-related complications, radiographic and functional healing at 6-8 weeks post-injury, length of stay in the emergency department, and facility charges. Comparisons between the two treatment groups (PEM and OP) will also be made with respect to each of these outcome variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pershad, MD, Study Director — University of Tennessee Health Sciences; Shehma Khan, MD, Principal Investigator — University of Tennessee Health Sciences
Locations (1):
- Lebonheur Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Background] Ward WT, Eberson CP, Otis SA, Wallace CD, Wellisch M, Warman JR, Leitch KK, Epps HR, Richards BS. Pediatric orthopaedic practice management: the role of midlevel providers. J Pediatr Orthop. 2008 Dec;28(8):795-8. doi: 10.1097/BPO.0b013e318183249f. No abstract available. PMID 19034167
- [Background] Ward WT, Rihn JA. Demographic and financial implications of pediatric emergency department fracture manipulation. J Pediatr Orthop. 2007 Dec;27(8):877-81. doi: 10.1097/BPO.0b013e3181558c4d. PMID 18209607
- [Background] Pershad J, Williams S, Wan J, Sawyer JR. Pediatric distal radial fractures treated by emergency physicians. J Emerg Med. 2009 Oct;37(3):341-4. doi: 10.1016/j.jemermed.2008.08.030. Epub 2009 Feb 6. PMID 19201136